CLINICAL TRIAL: NCT05501288
Title: Huashi Baidu Granule in the Treatment of Pediatric Patients With Mild Coronavirus Disease 2019: a Single-center, Open-label, Parallel-group Randomized Controlled Clinical Trial
Brief Title: Huashi Baidu Granule in the Treatment of Pediatric Patients With Mild Coronavirus Disease 2019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCMCIRB-K2022046-1
Record Dates: First submitted 2022-08-09; First posted 2022-08-15 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Coronavirus Disease 2019
Keywords: COVID-19; SARS-CoV-2; Omicron; Traditional Chinese Medicine; Clinical trial
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: randomly allocated 2:1 to receive oral HSBDG for 5 consecutive days (intervention group) and to receive compound pholcodine oral solution for 5 consecutive days (control group)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): receive oral HSBDG for 5 consecutive days
  Interventions: Drug: Huashi Baidu granule
- control group (Other): receive compound pholcodine oral solution for 5 consecutive days
  Interventions: Drug: compound pholcodine oral solution

INTERVENTIONS:
Drug: Huashi Baidu granule — Patients were given HSBDG the day after randomization, with a dose of 2.5g for age 3 to 6 years, 5 g for age 7 to 12 years, and 10 g for age 13 to 18 years, twice daily for 5 consecutive days.
  Arms: intervention group
Drug: compound pholcodine oral solution — Patients were given compound pholcodine oral solution (Bright Future Pharmaceuticals Factory, Hong Kong, CHN) the day after randomization, with a dose of 5 ml for age 3 to 6 years and 10 ml for age 7 to 18 years, three times daily for 5 consecutive days.
  Arms: control group

SUMMARY:
The investigators conducted a single-center, open-label, parallel-group randomized controlled trial to assess the efficacy and safety of a Chinese herb compound granule Huashi Baidu granule (HSBDG) in pediatric patients with laboratory-confirmed mild COVID-19. 108 recruited children (aged 3 to 18 years) with laboratory-confirmed mild COVID-19 were randomly allocated 2:1 to receive oral HSBDG for 5 consecutive days (intervention group) and to receive compound pholcodine oral solution for 5 consecutive days (control group). The negative conversion time of SARS-CoV-2 nucleic acid and symptom scores were recorded.

DETAILED DESCRIPTION:
This was a single-center, open-label, parallel-group randomized controlled clinical trial, with an allocation ratio of 2:1. Written consent was obtained from the parents of all participants. The study was conducted in accordance with the Declaration of Helsinki and the current Good Clinical Practice. The protocol was approved by the Institutional Ethics Committee of Shanghai Children's Medical Center (SCMCIRB-K2022046-1) Participants and setting Children who attended the COVID-19 Fangcang Shelter Hospitals in Shanghai, China, with laboratory-confirmed mild COVID-19 were screened for eligibility. The inclusion criteria were as follows: 1) compliance with the diagnostic criteria for mild COVID-19; 2) age 3 to 18 years. Participants who had underlying disease(s) such as chronic pulmonary disease, immunodeficiency, tumors, etc., allergy or intolerance to taking Chinese medicine herbs or compound pholcodine oral solution, or poor compliance (defined as inability to comply with the protocol) were excluded.

Sample size Two-sample T-tests allowing unequal variance were used for sample size calculation by Power Analysis and Sample Size Software 2021 (NCSS, LLC. Kaysville, Utah, USA). Group sample sizes of 64 and 32 achieve 85.0% power to reject the null hypothesis of equal means when the population mean difference is μ1 - μ2 = 10 - 11 = -1 with standard deviations of 1.42 for the intervention group and 1.56 for the control group, and with a significance level (alpha) of 0.05 using a two-sided two-sample unequal-variance t-test. The aim was to recruit 108 participants to allow for a 12% attrition rate.

Randomization and Blinding Patients were randomly assigned 2:1 to the intervention group or the control group by a researcher who was not otherwise involved in the study using random sequences generated by SPSS software 25.0 (IBM SPSS Statistics, Armonk, NY, USA). This was an open-label trial. Patients, investigators, and statisticians were not masked to the group assignment.

Intervention In the intervention group, patients were given HSBDG the day after randomization, with a dose of 2.5g for age 3 to 6 years, 5 g for age 7 to 12 years, and 10 g for age 13 to 18 years, twice daily for 5 consecutive days. In the control group, patients were given compound pholcodine oral solution (Bright Future Pharmaceuticals Factory, Hong Kong, CHN) the day after randomization, with a dose of 5 ml for age 3 to 6 years and 10 ml for age 7 to 18 years, three times daily for 5 consecutive days. The day of randomization was set as day 0. By free Instant messaging software (WeChat; Tencent, Shenzhen, CHN) available on smart phones, parents received questionnaires (Table S1 for symptom scores at days 0, 3 and 5) and be asked to complete them truthfully. For each patient, one SARS-CoV-2 nucleic acid real-time PCR test for the specimen from the upper respiratory tract was performed daily. Patients would be not considered to be discharged until two consecutive negative reports were confirmed.

Primary outcome The primary outcome of the study was the time for SARS-CoV-2 nucleic acid negative conversion after randomization. The time from day 0 to the day of two consecutive negative reports confirmed was defined as the negative conversion time.

Secondary outcomes The secondary outcomes for the study were symptom improvements at days 3 and 5, and antibiotic use and side effects from day 1 to discharge. Total symptom score was the sum of the scores of primary symptoms (fever, cough, expectoration, sore throat, wheezing, and chest pain) and secondary symptoms (dry stool, dark urine or oliguria, poor appetite, low energy, tired, nausea or vomiting, and diarrhea).

Statistical analysis Data were presented as frequencies and percentages for categorical variables and as medians and interquartile range (IQR) for continuous variables. Categorical variables were compared by the chi-square test. Continuous variable comparisons were performed by the Mann-Whitney U test. P-value < 0.05 was considered to be statistical significance. All analyses were performed using SPSS software 25.0 (IBM SPSS Statistics, Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* attend the COVID-19 Fangcang Shelter Hospitals in Shanghai, China
* with laboratory-confirmed COVID-19
* compliance with the diagnostic criteria for mild COVID-19
* age 3 to 18 years.

Exclusion Criteria:

* with underlying disease(s) such as chronic pulmonary disease, immunodeficiency, tumors, etc.,
* allergy or intolerance to taking Chinese medicine herbs or compound pholcodine oral solution
* with poor compliance (defined as inability to comply with the protocol)
* decline to participate

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Time for SARS-CoV-2 nucleic acid negative conversion | up to three weeks
  The primary outcome of the study was the time for SARS-CoV-2 nucleic acid negative conversion after randomization. The time from day 0 to the day of two consecutive negative reports confirmed was defined as the negative conversion time.

SECONDARY OUTCOMES:
Symptom score, antibiotic use, and side effects | up to three weeks
  The secondary outcomes for the study were symptom scores on days 3 and 5, and antibiotic use and side effects from day 1 to discharge. Total symptom score was the sum of the scores of primary symptoms (fever, cough, expectoration, sore throat, wheezing, and chest pain) and secondary symptoms (dry stool, dark urine or oliguria, poor appetite, low energy, tired, nausea or vomiting, and diarrhea). For each primary symptom, no problem, minor problem, moderate problem, and major problem correspond to 0, 2, 4, and 6 points, respectively. For each secondary symptom, no problem, minor problem, moderate problem, and major problem correspond to 0, 1, 2, and 3 points, respectively. The total score is 0 to 60. The higher the score, the more serious the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Gao, MD, Principal Investigator — Shanghai Children's Medical Center; Yong Yin, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai children's medical center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data are available from the corresponding author upon reasonable request.